CLINICAL TRIAL: NCT07352813
Title: A Comparative Evaluation of the Clinical Effectiveness of Computer-Assisted Intraosseous and Infiltration Anesthesia Techniques in Children With Molar-Incisor Hypomineralization
Brief Title: Intraosseous vs Infiltration Anesthesia in Molar-Incisor Hypomineralization (MIH) Children
Acronym: MIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Gülsevim ODA, Asst. Prof., Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EK-2025-263
Record Dates: First submitted 2025-12-18; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Molar Incisor Hypomineralization; Hypersensitivity
Keywords: caries; dental anxiety; dental pain; molar incisor hypomineralization
MeSH Terms: conditions — Molar Hypomineralization; Hypersensitivity; Toothache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraosseous Anesthesia (Experimental): The intraosseous anesthesia technique will be administered using the computer-assisted anesthesia device (SleeperOne® 5) and applied to either the right or left upper permanent molar, assigned at random.
  Interventions: Procedure: Intraosseous anaesthesia using a computerized system
- Infiltration Anesthesia (Active Comparator): The infiltration anesthesia technique will be administered using the SleeperOne® 5 device and applied to the opposite side of the same patient.
  Interventions: Procedure: Infiltration anaesthesia using a computerized system

INTERVENTIONS:
Procedure: Intraosseous anaesthesia using a computerized system — Articaine hydrochloride: 40 mg/mL Epinephrine (adrenaline): 0.012 mg/mL, corresponding to a 1:100,000 dilution.
  Arms: Intraosseous Anesthesia
Procedure: Infiltration anaesthesia using a computerized system — Articaine hydrochloride: 40 mg/mL Epinephrine (adrenaline): 0.012 mg/mL, corresponding to a 1:100,000 dilution.
  Arms: Infiltration Anesthesia

SUMMARY:
This study aims to compare the effectiveness of intraosseous and infiltration anesthesia techniques administered using a computer-assisted anesthesia device (SleeperOne® 5; Dental HiTec, France) during restorative treatments of permanent first molars affected by Molar-Incisor Hypomineralization (MIH) in children. Clinical effectiveness will be evaluated based on the Visual Analogue Scale (VAS), behavioral pain response, pulse rate , salivary chromogranin A levels, and the need for additional anesthesia.

DETAILED DESCRIPTION:
Children who present to the Pediatric Dentistry Clinic of Ankara Yıldırım Beyazıt University, Dental Research and Application Center, and are deemed eligible for inclusion in the study based on routine clinical examination and radiographic evaluation, will be provided with written and verbal information regarding the purpose and scope of the research. Informed consent will be obtained from those children and their legal guardians who voluntarily agree to participate in the study.

The study plans to include 30 children aged between 6 and 12 years, who have no systemic diseases and present with Molar-Incisor Hypomineralization (MIH) and carious lesions not extending to the pulp tissue in their maxillary permanent first molars.

A three-session treatment protocol will be administered to participants who meet the inclusion criteria and have signed the informed consent form. A minimum interval of one week will be maintained between sessions, and the sequence of interventions will be determined through randomization.

First Session:

In the first session, a detailed medical and dental history of the patient will be obtained. During the intraoral examination, teeth affected by MIH will be identified, and the degree of MIH as well as the presence of carious lesions will be evaluated through clinical and radiographic examination. All findings will be recorded in the patient data form.

In this session, no invasive procedures will be performed. The materials and methods to be used will be explained to the patient, and the Frankl Behavior Rating Scale will be applied to determine the preoperative anxiety level, serving as an acclimatization session.

Second Session:

The anesthesia method to be applied to the patient's upper right first permanent molar (tooth no. 16) in the second session will be determined using a randomization method. Before the administration of anesthesia, the technique of the procedure will be explained verbally to the pediatric patient; the first saliva sample will be collected, and pulse rate values will be measured and recorded using a pulse oximeter. The anesthesia method determined by randomization will be applied to tooth number 16. During anesthesia administration, the patient will be asked to evaluate the pain level experienced using the Visual Analogue Scale (VAS) (0 = no pain, 10 = unbearable pain). After anesthesia, the pulse rate will again be recorded, and the second saliva sample will be collected. The carious tissue of the affected tooth will be removed using a high-speed and low-speed handpiece. At this stage, the heart rate will also be measured and recorded using the pulse oximeter. At the end of the treatment, the third saliva sample will be collected, and the patient will be asked to evaluate the pain level experienced using the VAS. Saliva samples as well as immediately after treatment completion and stored at -20 °C until biochemical analysis.

Throughout the treatment, the patient's behavioral responses will be video recorded and objectively evaluated by an independent observer, blinded to the anesthesia method, using the FLACC scale. The need for additional anesthesia and the efficacy of the anesthesia will be assessed after treatment.

Third Session:

In the third session, the anesthesia technique will be changed, and anesthesia will be administered to the contralateral first molar tooth (in the symmetrical arch) with the same indication. The procedures performed in the second session will be repeated.

At the conclusion of this study, the comparison of anesthesia techniques used in the treatment of MIH-affected teeth in children will enable the identification of a minimally invasive and effective approach to anesthesia. It is well established that teeth affected by MIH exhibit an altered response to anesthesia due to hypersensitivity and structural changes in the enamel. This study aims to contribute to the existing gap in the scientific literature on this topic. The comparative evaluation of computer-assisted intraosseous and infiltration anesthesia techniques will facilitate evidence-based decision-making in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals applying to the Department of Pedodontics, Ankara Yıldırım Beyazıt University Faculty of Dentistry,
* Systemically healthy individuals,
* Individuals without any known allergies,
* Children between the ages of 6 and 12 years,
* Scoring 3-4 according to the Frankl Behavior Rating Scale,
* Children and their legal guardians who, after reading and listening to the informed consent form, fully understand its content and voluntarily provide both verbal and written consent,
* Children with contralateral and homologous maxillary first permanent molars affected by molar-incisor hypomineralization (MIH) and scoring 3-4 according to the MIH Treatment Need Index criteria,
* Children with no emergency treatment needs, such as dental pain,
* Both male and female volunteers.

Exclusion Criteria:

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-11-07 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Salivary Chromogranin A Levels | During dental treatment (Day 1): Baseline (before local anesthesia administration) Immediately after local anesthesia application Immediately after completion of the restorative procedure
  To objectively assess the stress levels experienced by children during dental treatment, changes in salivary chromogranin A concentrations will be measured at predefined time points during the procedure.

SECONDARY OUTCOMES:
Pulse Rate | During dental treatment (Day 1): • Baseline (before local anesthesia administration) • Immediately after local anesthesia application • Throughout the restorative treatment procedure
  Patients' heart rates will be measured using a pulse oximeter to assess physiological stress responses during dental treatment.
Visual Analogue Scale [VAS] | During dental treatment (Day 1): Immediately after local anesthesia application Immediately after completion of the restorative procedure
  The Visual Analogue Scale (VAS) will be used to assess perceived pain intensity during dental treatment. VAS is a validated and widely used psychometric instrument for quantifying subjective pain experience on a 10-point scale, ranging from "No pain" to "Unbearable pain."
Behavioral Pain Response (FLACC Score): | TDuring dental treatment (Day 1): Throughout the restorative treatment procedure (single assessment)
  Behavioral pain response will be assessed using the FLACC scale, which consists of five behavioral categories: Face, Legs, Activity, Cry, and Consolability. Each category is scored from 0 to 2, yielding a total score ranging from 0 to 10.
  During the restorative procedure, video recordings will be obtained. An independent observer (E.Ü.A.), blinded to the anesthesia method, will evaluate the recordings and score the child's behavioral responses using the FLACC scale.
Need for Additional Anesthesia | During dental treatment (Day 1): Throughout the treatment procedure (single assessment)
  The adequacy of the administered anesthesia during dental treatment will be evaluated by the researcher. The requirement for additional anesthesia will be recorded as a dichotomous outcome (yes/no).
Anesthesia Efficacy Assessment (Efficacy Scale): | Periprocedural (Day 1; immediately after completion of the restorative procedure)
  Anesthesia efficacy will be assessed using an efficacy scale that evaluates the clinical success of the administered anesthesia based on the presence or absence of pain during the dental procedure. This scale reflects both the patient's pain experience and the clinician's ability to complete the planned treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe I Cihan, Professor, Study Chair — Ankara Yıldırım Beyazit University Faculty of Dentistry
Locations (1):
- Ankara Yıldırım Beyazıt University Faculty of Dentistry, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Dixit UB, Joshi AV. Efficacy of Intraosseous Local Anesthesia for Restorative Procedures in Molar Incisor Hypomineralization-Affected Teeth in Children. Contemp Clin Dent. 2018 Sep;9(Suppl 2):S272-S277. doi: 10.4103/ccd.ccd_252_18. PMID 30294157
- [Background] Cabasse C, Marie-Cousin A, Huet A, Sixou JL. Computer-assisted intraosseous anaesthesia for molar and incisor hypomineralisation teeth. A preliminary study. Odontostomatol Trop. 2015 Mar;38(149):5-9. PMID 26058304
- [Background] Berrendero S, Hriptulova O, Salido MP, Martinez-Rus F, Pradies G. "Comparative study of conventional anesthesia technique versus computerized system anesthesia: a randomized clinical trial". Clin Oral Investig. 2021 Apr;25(4):2307-2315. doi: 10.1007/s00784-020-03553-5. Epub 2020 Aug 29. PMID 32862249
- [Background] Rhaiem M, Chatti M, Elelmi Y, Ben Haj Khalifa A, Masmoudi F, Baaziz A. Effective anaesthesia when treating teeth affected by molar incisor hypomineralisation (MIH): a systematic review. Eur Arch Paediatr Dent. 2025 Oct;26(5):861-876. doi: 10.1007/s40368-025-01057-y. Epub 2025 May 30. PMID 40445534